CLINICAL TRIAL: NCT06569225
Title: Perioperative Therapy With Gemcitabine/Cisplatin/Nab-Paclitaxel and Rilvegostomig for Patients With Resectable Intrahepatic Cholangiocarcinoma (iCCA) - A Phase II Trial
Brief Title: Gemcitabine/Cisplatin/Nab-Paclitaxel and Rilvegostomig in Resectable iCCA
Acronym: NEOLANGIO
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University Health Network, Toronto (Other)
Collaborators: Sunnybrook Health Sciences Centre (Other); Hamilton Health Sciences Corporation (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 24-5716
Record Dates: First submitted 2024-08-21; First posted 2024-08-26 (Actual); Last update posted 2024-08-26 (Actual); Status verified 2024-08

CONDITIONS: Cholangiocarcinoma Resectable
Keywords: CCA; Biliary cancer; Neo-adjuvant and adjuvant therapy
MeSH Terms: conditions — Biliary Tract Neoplasms | interventions — Gemcitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Gemcitabine/Cisplatin/Nab-Paclitaxel and Rilvegostomig (Experimental)
  Interventions: Drug: Gemcitabine/Cisplatin/Nab-Paclitaxel and Rilvegostomig

INTERVENTIONS:
Drug: Gemcitabine/Cisplatin/Nab-Paclitaxel and Rilvegostomig — : Patients will receive prior to surgery: 2 cycles of combinational therapy with Gemcitabine (800mg) /Cisplatin (25mg) /Nab-Paclitaxel (100mg) and Rilvegostomig (Q3W). Post-surgical resection, adjuvant therapy will consist of 4 cycles of Gemcitabine (1000mg) /Cisplatin (25mg) and Rilvegostomig (Q3W). Rilvegostomig (Q3W) will be continued for a total of 12 months in the adjuvant phase

SUMMARY:
Biliary tract cancer is a highly aggressive and heterogeneous group of gastrointestinal cancers that arise from the intra- or extrahepatic bile ducts (CCA), or the gallbladder (GBC)(1-3). While it accounts for only 0.7% of all malignant tumors and 3% of all gastrointestinal malignancies in adults, both incidence and mortality are increasing. Biliary tract cancers usually present at an advanced stage, with only approximately 20% of patients being diagnosed with an early-stage disease (1, 2, 4). There is a high risk of recurrence post curative radical resection, with 60-70% of patients recurring within 5 years, with 5-year survival of around 25% (1, 2, 5). There is evidence for use of adjuvant chemotherapy with fluoropyrimidine- based regimens as per the BILCAP and ASCOT phase III trials [(5-7).However, despite advances in adjuvant treatment, recurrence rates after resection of BTC remain high even with adjuvant chemotherapy. For example, in the BILCAP study, 5-year RFS was reported as 33.9% (95% CI: 27.6 to 40.2) (1). Therefore, an unmet need exists to optimize peri-operative treatment to reduce recurrence and improve outcomes in patients with resectable BTC.

DETAILED DESCRIPTION:
The only curative management for iCCA is radical surgical resection. However, less than 35% of patients present with resectable disease at diagnosis, and postoperative recurrence and relapse rates are around 50-70%. Despite advances in diagnostics and therapeutic interventions, prognosis remains poor with an overall 5-year survival of less than 20%.1

The results of the TOPAZ-12 and KEYNOTE-9663 study have established PD-L1 (durvalumab) and PD-1 (pembrolizumab) inhibition in combination with gemcitabine and cisplatin as a new standard of care highlighting the role of immune checkpoint inhibition in advanced biliary tract cancer (BTC). In addition, the combination of Nab-Paclitaxel and gemcitabine, cisplatin has demonstrated efficacy in advanced BTC4. Several clinical trials evaluating the efficacy of neoadjuvant combinational therapy with gemcitabine, cisplatin and PD-L1 inhibition are ongoing (NCT04989218, NCT06050252, NCT04308174). Neoadjuvant treatment in iCCA allows for delivery of treatment pre surgery and can induce pathological responses and thereby improve survival. Rilvegostomig is a novel anti-TIGIT/anti-PD-1 bispecific antibody that is currently investigated in a Phase I/II clinical trial (ARTEMIDE-01, NCT04995523) for advanced or metastatic PD-L1-positive non-small cell lung cancer. The study provided promising preliminary evidence on the safety and efficacy of Rilvegostomig.5,6 Furthermore, a Phase III clinical trial (ARTEMIDE-Biliary01) using Rilvegostomig in combination with Capecitabine or Gemcitabine/Cisplatin or S-1 as adjuvant therapy for BTC after resection is underway. The efficacy of Gemcitabine/Cisplatin/Nab-Paclitaxel and Rilvegostomig as neoadjuvant treatment in resectable iCCA has yet to be established.

This is a phase II, open-label multi-centre study to assess efficacy of Gemcitabine/Cisplatin/Nab-Paclitaxel and Rilvegostomig treatment in pre-surgical setting for upfront resectable iCCA, followed by adjuvant Gemcitabine/Cisplatin and Rilvegostomig.

40 patients are expected to enrol with resectable iCCA at three sites. Patients will receive prior to surgery: 2 cycles of combinational therapy with Gemcitabine (800mg) /Cisplatin (25mg) /Nab-Paclitaxel (100mg) and Rilvegostomig (Q3W). Post-surgical resection, adjuvant therapy will consist of 4 cycles of Gemcitabine (1000mg) /Cisplatin (25mg) and Rilvegostomig (Q3W). Rilvegostomig (Q3W) will be continued for a total of 12 months in the adjuvant phase.

All participants will be followed for survival until the end of study.

Dosing of Gemcitabine/Cisplatin/Nab-Paclitaxel and Rilvegostomig may be delayed per the trial management group's discretion but dose reduction will not be allowed. Toxicity management for Gemcitabine/Cisplatin/Nab-Paclitaxel and Rilvegostomig-related toxicity, including management of immune-mediated reactions, infusion-related reactions, and non-immune-mediated reactions will be provided in the Toxicity Management Guidelines

ELIGIBILITY:
Inclusion Criteria:

1. Patient must be capable of providing written informed consent.
2. Age >18 years at time of study entry
3. Histologically proven intrahepatic cholangiocarcinoma
4. Complete surgical resection of the tumor must be achievable*. Resection should include a portal lymphadenectomy as per standard of care.
5. No prior cytotoxic, targeted or immune therapy
6. Have provided archival tumor tissue sample or preferably freshly obtained biopsy of a tumor lesion not previously irradiated for mandatory pre-treatment evaluation (baseline).
7. Eastern Cooperative Oncology Group (ECOG) performance status (PS) of 0 or 1
8. Estimated life expectancy >3 months
9. Exclusion of distant metastases by CT or MRI of abdomen, pelvis, and thorax, bone scan or MRI (if bone metastases are suspected due to clinical signs). Exclusion of the infiltration of any adjacent organs or structures by CT or MRI, indicating an unresectable situation
10. If underlying liver cirrhosis, Childs Pugh score of 5 or 6
11. If underlying liver disease, ALBI grade ≤2†
12. Patients with HBV infection, which is characterized by positive hepatitis B surface antigen (HBsAg) and/or hepatitis B core antibodies (anti-HBcAb) with detectable HBV DNA (≥10 IU/ml or above the limit of detection per local lab standard), must be treated with antiviral therapy, as per institutional practice, to ensure adequate viral suppression (HBV DNA ≤2000 IU/mL) prior to study entry. Patients must remain on antiviral therapy for the study duration and for 6 months after the last dose of study medication. Patients who test positive for anti-hepatitis B core (HBc) with undetectable HBV DNA (<10 IU/ml or under limit of detection per local lab standard) do not require anti-viral therapy prior to study entry. These subjects will be tested at every cycle to monitor HBV DNA levels and initiate antiviral therapy if HBV DNA is detected (≥10 IU/ml or above the limit of detection per local lab standard). HBV DNA detectable subjects must initiate and remain on antiviral therapy for the study duration and for 6 months after the last dose of study medication.
13. Patients with HCV infection must have management of this disease per local institutional practice throughout the study. HCV diagnosis is characterized by the presence of detectable HCV ribonucleic acid (RNA) or anti-HCV antibody upon enrollment.
14. Evidence of post-menopausal status or negative serum pregnancy test for female pre-menopausal patients.
15. Adequate normal organ and marrow function as defined below within screening period:

    * Haemoglobin ≥9.0 g/dL
    * Absolute neutrophil count (ANC ≥1.0 × 109 /L)
    * Platelet count ≥100 × 109/L
    * Serum bilirubin ≤1.5 x institutional upper limit of normal (ULN). <<This will not apply to patients with confirmed Gilbert's syndrome (persistent or recurrent hyperbilirubinemia that is predominantly unconjugated in the absence of hemolysis or hepatic pathology), who will be allowed only in consultation with their physician.
    * AST (SGOT)/ALT (SGPT) ≤5 x institutional upper limit of normal.
    * Measured creatinine clearance (CL) >50 mL/min or Calculated creatinine clearance

    CL>50 mL/min by the Cockcroft-Gault formula (Cockcroft and Gault 1976) or by 24-hour urine collection for determination of creatinine clearance:

    Males:

    Creatinine CL (mL/min) = Weight (kg) x (140 - Age) 72 x serum creatinine (mg/dL)

    Females:

    Creatinine CL (mL/min) = Weight (kg) x (140 - Age) x 0.85 72 x serum creatinine (mg/dL)
    * Albumin ≥2.8g/dl
    * International normalized ratio ≤1.5 (for patients receiving Warfarin, please consult with the study physician)
16. Patient is willing and able to comply with the protocol for the duration of the study including undergoing treatment and scheduled visits and examinations including follow up.

    * Resectability is at the discretion of the investigators at each site but must be discussed at a multidisciplinary tumour board.

      * based on albumin and bilirubin; ALBI score = (log10 bilirubin [umol/L] x0.66) + (albumin [g/L] x -0.0852). ALBI grade 1= score ≤ -2.60.

Exclusion Criteria:

Patients should not enter the study if any of the following exclusion criteria are fulfilled at time of study enrolment or where indicated:

1. Locally unresectable tumor or metastatic disease:

   1. Radiological evidence suggesting inability to resect with curative intent whilst maintaining adequate vascular inflow and outflow
   2. Radiological evidence of direct invasion into adjacent organs.
   3. Radiological evidence of extrahepatic metastatic disease (except regional lymph nodes - stations 9 and 12
2. Contraindication to any of the study drugs
3. Any concurrent chemotherapy, investigational product, biologic or hormonal therapy for cancer treatment
4. Are currently participating in or has participated in a study of an investigational agent or has used an investigational device within 4 weeks or for a period of at least 5 half-lives of the respective drug/IMP (whichever is longer) before screening and during Screening for this trial.
5. Have a diagnosis of immunodeficiency or are receiving chronic systemic steroid therapy (in dosing exceeding 10 mg daily of prednisone equivalent) or any other form of immunosuppressive therapy within 7 days prior to the first dose of study drug.
6. Have a known additional malignancy that is progressing or has required active treatment within the past 2 years.

   Note: Participants with basal cell carcinoma of the skin, squamous cell carcinoma of the skin or carcinoma in situ (e.g., breast carcinoma, cervical cancer in situ) that have undergone potentially curative therapy are not excluded.
7. Have active autoimmune disease that has required systemic treatment in the past 2 years (i.e., with use of disease modifying agents, corticosteroids or immunosuppressive drugs). Replacement therapy (e.g., thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc.) is not considered a form of systemic treatment and is allowed.
8. Have a history of (non-infectious) pneumonitis/interstitial lung disease that required steroids or has current pneumonitis/interstitial lung disease.
9. Have an active infection requiring systemic therapy (exception: HBV and HCV infection).
10. Have a history of Human Immunodeficiency Virus (HIV) (mandatory testing for HIV during screening is required).
11. Have known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial.
12. Female patients who are pregnant or breastfeeding or male or female patients of reproductive potential who are not willing to employ highly effective birth control from screening to 6 months after the last dose of study treatment. Not engaging in sexual activity, per the patient's preferred and usual lifestyle, for the total duration of the treatment and 6 months after the last dose of study treatment is an acceptable practice.

    Note: Females of childbearing potential are defined as those who are not surgically sterile (ie, bilateral salpingectomy, bilateral oophorectomy, or complete hysterectomy) or not post menopausal.

    Women will be considered post-menopausal if they have been amenorrheic for 12 months without an alternative medical cause. The following age-specific requirements apply:
    * Women <50 years of age would be considered post-menopausal if they have been amenorrheic for 12 months or more following cessation of exogenous hormonal treatments and if they have luteinizing hormone and follicle-stimulating hormone levels in the post-menopausal range for the institution.
    * Women ≥50 years of age would be considered post-menopausal if they have been amenorrheic for 12 months or more following cessation of all exogenous hormonal treatments, had radiation-induced menopause with last menses >1 year ago, or had chemotherapy-induced menopause with last menses >1 year ago.
    * Women who are surgically sterile (i.e., bilateral salpingectomy, bilateral oophorectomy, or complete hysterectomy) are eligible.

    Highly effective methods of contraception, defined as one that results in a low failure rate (i.e., less than 1% per year) when used consistently and correctly. Note that some contraception methods are not considered highly effective (e.g., male or female condom with or without spermicide; female cap, diaphragm, or sponge with or without spermicide; non copper containing intrauterine device; progestogen-only oral hormonal contraceptive pills where inhibition of ovulation is not the primary mode of action [excluding Cerazette/desogestrel, which is considered highly effective]; and triphasic combined oral contraceptive pills). Serum levels of contraceptive hormones may be altered by concomitant use of other drugs. Therefore, drug interactions should always be considered when prescribing hormonal contraception; there could be a risk of contraceptive failure or other adverse effects.
13. Legal incapacity or limited legal capacity.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2024-12-15 (Estimated); Primary Completion 2027-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Major pathological response (MPR), defined as >70% tumor necrosis | 2 years
  To determine pathological response rate to neoadjuvant Gemcitabine/Cisplatin/Nab-Paclitaxel and Rilvegostomig in resected tumour

SECONDARY OUTCOMES:
Objective response rate (ORR) | 3 years
  To determine the radiologic objective response rate (ORR) to neoadjuvant Gemcitabine/Cisplatin/Nab-Paclitaxel and Rilvegostomig.
The number of patients who experience a surgical delay and/or drop off due to treatment related adverse events (TRAEs) or progressive disease | 2 years
  To assess feasibility of pre-operative treatment of Gemcitabine/Cisplatin/Nab-Paclitaxel and Rilvegostomig
The number of ≥ grade 3 adverse events (AEs) or immune related adverse events that occur during treatment | 3 years
  To assess safety of pre-operative treatment with Gemcitabine/Cisplatin/Nab-Paclitaxel and Rilvegostomig.
Rate of R0 | 2 years
  Number of resections with negative margins

CONTACTS AND LOCATIONS:
Locations (1):
- University Health Network, Toronto General Hospital, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Undecided